CLINICAL TRIAL: NCT00656929
Title: A Randomized Controlled Trial of Vitamin D3 Supplementation for the Prevention of Viral Upper Respiratory Tract Infections
Brief Title: Randomized Controlled Trial of Vitamin D3 Supplementation for Viral Upper Respiratory Tract Infections (URI) Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Responsible Party: John F. Aloia, M.D., Winthrop University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WUH06034
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Viral Upper Respiratory Tract Infection
Keywords: Vitamin D; Viral URI; Influenza; Colds
MeSH Terms: conditions — Influenza, Human | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Vitamin D3 50 mcg (2000 IU) daily
  Interventions: Dietary Supplement: Vitamin D3
- 2 (Placebo Comparator): Placebo tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 (cholecalciferol) 50 mcg (2000 IU) daily x 3 months
  Other Names: cholecalciferol
  Arms: 1
Other: Placebo — Placebo tablets
  Arms: 2

SUMMARY:
Background: Vitamin D has been shown to be an important immune system regulator. Vitamin D insufficiency during the winter may cause increased susceptibility to infections, particularly viral upper respiratory tract infections (URIs).

Objective: To determine whether vitamin D supplementation during the winter season prevents or decreases URI symptoms in adults.

Methods: A randomized, double-blind, placebo-controlled trial was conducted in 162 adults. Participants were randomized to receive vitamin D3 50 mcg (2000 IU) daily or matching placebo for 12 weeks from December 2006 to March 2007. A biweekly questionnaire was used to record the incidence and severity of URI symptoms

ELIGIBILITY:
Inclusion Criteria:

* ambulatory adult age 18-80 and stable medical condition with no change in medications for 6 months prior to study entry.

Exclusion Criteria:

* morbid obesity (body mass index > 35 kg/m2)
* current tobacco use
* history of hypercalcemia, nephrolithiasis or sarcoidosis
* pregnancy
* recent hospitalization
* current liver or kidney disorders, malignancy and malabsorption
* use of immunosuppressants or medications that interfere with vitamin D metabolism such as phenytoin and carbamazepine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2006-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To see whether vitamin D3 supplementation during the winter prevents viral URI. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John F Aloia, MD, Principal Investigator — Winthrop University Hospital